CLINICAL TRIAL: NCT02131480
Title: A Multicentric Phase II Trial Studying Efficacy of Doxorubicin Associated With Trabectedin (Yondelis) in First Line Treatment on Patients With Metastatic Leiomyosarcoma (Uterus or Soft Tissue) and/or Inoperable Relapse
Brief Title: Study of Doxorubicin and Trabectedin in First Line Treatment on Patients With Metastatic Leiomyosarcoma
Acronym: LMS02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-012430-70; 2008/1485 (Other: CSET number)
Record Dates: First submitted 2014-05-05; First posted 2014-05-06 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Uterus Leiomyosarcoma; Soft Tissue Leiomyosarcoma
MeSH Terms: interventions — Doxorubicin; Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soft tissue (Experimental)
  Interventions: Drug: Doxorubicin; Drug: Trabectedin
- Uterus (Experimental)
  Interventions: Drug: Doxorubicin; Drug: Trabectedin

INTERVENTIONS:
Drug: Doxorubicin — 60 mg/m²
  Other Names: Adriamycin
Drug: Trabectedin — 1,1 mg/m²
  Other Names: Yondelis®

SUMMARY:
Uterine leiomyosarcomas and soft tissues are rare tumors with a poor prognosis when metastatic or locally advanced. They have an average chemosensitivity mainly to doxorubicin, ifosfamide, cisplatin, gemcitabine and trabectedin but response rates in combination in first line does not exceed 55% for uterine leiomyosarcomas and 35% for leiomyosarcomas of soft tissue.

The trabectedin is a new cancer drug that has obtained marketing authorization after failure of anthracyclines and ifosfamide in the treatment of soft tissue sarcomas (STM) in Europe. It has especially shown efficacy in myxoid liposarcomas, leiomyosarcomas and synoviosarcoma.

This study aims to evaluate the usefulness of the combination of trabectedin with doxorubicin in first-line treatment of uterine or soft tissue leiomyosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic leiomyosarcoma (uterus or soft tissue) in inoperable relapse with no previous chemotherapy
* At least one measurable lesion according to RECIST criteria before inclusion. At least one of the target is in a none irradiated area
* Aged >/= 18 years and physiological age </= 70 years
* PS </= 2
* Normal hematological function (Polymorphonuclear Neutrophils >/= 1500/mm3, platelets >/= 100 000/mm3)
* Normal kidney function (creatinine < 1.5xN)
* Creatinine phosphokinase </= 2.5xN
* Normal hepatic function (total bilirubin </= 1xN; transaminase </= 2.5xN and alkaline phosphatase </= 1.5xN)
* Cardiac function: normal echography and/or isotopic ventriculography (FR>30%, FEVG > 50%)
* Patients able to procreate must use a birth control device during treatment and during 3 months after treatment for women; 5 months for men
* Signed informed consent
* Patient under affiliated to a system of care

Exclusion Criteria:

* Any other histological type of uterus sarcoma (carcinosarcoma...) or soft tissue
* Specific contraindication to the treatment
* Previous or evolutive mental disease
* Previous cancer
* Symptomatic or known brain metastasis
* Previous radiotherapy ont he only measurable lesion
* Previous allograft or autograft
* Known positive serology (HIV, HbC, HbS)
* Pregnant or breastfeeding women
* Impossibility to follow the treatment for geographical, social or mental reason
* Patients under legal protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Disease control rate | Assessed every 6 weeks from inclusion up to 6 months
  Disease control rate (objective response + stability) as defined by RECIST criteria

SECONDARY OUTCOMES:
Response rate | Assessed every 6 weeks from inclusion up to 6 months
  Assessed using RECIST criteria
Progression Free Survival | Assessed every 6 weeks from inclusion up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Pautier P, Floquet A, Chevreau C, Penel N, Guillemet C, Delcambre C, Cupissol D, Selle F, Isambert N, Piperno-Neumann S, Saada-Bouzid E, Bertucci F, Bompas E, Alexandre J, Collard O, Lebrun-Ly V, Soulier P, Toulmonde M, Le Cesne A, Lacas B, Duffaud F; French Sarcoma Group. A single-arm multicentre phase II trial of doxorubicin in combination with trabectedin in the first-line treatment for leiomyosarcoma with long-term follow-up and impact of cytoreductive surgery. ESMO Open. 2021 Aug;6(4):100209. doi: 10.1016/j.esmoop.2021.100209. Epub 2021 Jul 26. PMID 34325109
- [Derived] Pautier P, Floquet A, Chevreau C, Penel N, Guillemet C, Delcambre C, Cupissol D, Selle F, Isambert N, Piperno-Neumann S, Thyss A, Bertucci F, Bompas E, Alexandre J, Collard O, Lavau-Denes S, Soulie P, Toulmonde M, Le Cesne A, Lacas B, Duffaud F; French Sarcoma Group. Trabectedin in combination with doxorubicin for first-line treatment of advanced uterine or soft-tissue leiomyosarcoma (LMS-02): a non-randomised, multicentre, phase 2 trial. Lancet Oncol. 2015 Apr;16(4):457-64. doi: 10.1016/S1470-2045(15)70070-7. Epub 2015 Mar 18. PMID 25795402